CLINICAL TRIAL: NCT05273060
Title: Regenerative Medicine Approach to Nasal Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brittany E. Howard, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-004941
Record Dates: First submitted 2022-01-09; First posted 2022-03-10 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Nasal Surgical Procedures; Regenerative Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Nasal Reconstruction Planning (No Intervention): Subjects undergoing nasal reconstruction will have standard planning for procedure.
- 3D Nasal Reconstruction Planning (Experimental): Subjects undergoing nasal reconstruction will have 3D planning utilized by the surgical team for the procedure.
  Interventions: Procedure: 3D Nasal Reconstruction Planning

INTERVENTIONS:
Procedure: 3D Nasal Reconstruction Planning — 3D molds or models to use in the reconstruction of nasal cartilage
  Arms: 3D Nasal Reconstruction Planning

SUMMARY:
The purpose of this study is to gather information on the safety and effectiveness and compare nasal reconstruction standard planning versus 3D preoperative scanning/printing/planning.

DETAILED DESCRIPTION:
Patients with nasal defects from cancer, trauma, prior surgery, or birth often require complex reconstruction. Current techniques involve hand sketched skin templates and/or hand carved cartilage grafts that are formed intraoperatively for nasal reconstruction. This process is time consuming, heavily depends on the surgeon's skill, cannot be standardized, and is difficult to visualize with patients preoperatively. To overcome these barriers and shift surgical paradigms, we will use a regenerative medicine approach to nasal reconstruction to create patient specific and individualized results. We will leverage regenerative medicine techniques of 3D surface mapping, 3D printing and modeling, and new tissue preparation techniques for skin template creation and sculpting of cartilage grafting. Clinically this will improve patient specific outcomes, increase reproducibility, reduce operative times, and allow for an individualized approach to nasal reconstruction. This will be achieved by (1) establishing ideal diced cartilage graft parameters in the laboratory setting for moldable cartilage graft formation. This knowledge will be applied to (2) create diced cartilage grafts for nasal dorsum and tip reconstruction from 3D printed nasal molds. For nasal skin reconstruction, (3) 3D facial scans of patients' preoperatively will be used to generate patient specific templates for skin reconstruction. Ultimately, (4) these regenerative medicine techniques of cartilage and skin reconstruction performed with 3D planning can be shared in an interactive format with patients preoperatively. This will allow patients to be involved in the surgical planning of their nasal reconstruction to increase their autonomy and the individualization of their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males or female, age range is ≥ 18 to ≤ 100, based on historical surgical experience.
* Patients undergoing nasal reconstruction.
* Patients will be identified from the Facial Plastic Surgery clinic of the PI.

Exclusion Criteria:

- Patients < 18 are excluded because these cases are in combination with providers from PCH and patients have shared/limited postoperative follow up as a result.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Viable nasal reconstruction | 6 months
  Total number of subjects to have successful nasal reconstruction with transfer of viable tissue to reconstruct nasal defect

SECONDARY OUTCOMES:
Nasal breathing | 6 months
  Total number of subjects to have ability to move air through the nose for purposes of breathing

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Howard, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No